CLINICAL TRIAL: NCT06656715
Title: Symptom Burden and Health Related Quality of Life of Cancer Patients With Concurrent Heart Failure
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1125
Record Dates: First submitted 2024-10-11; First posted 2024-10-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SingleArm: Symptom Assessment and Comparison

SUMMARY:
To describe and compare the symptom burden in cancer patients with concurrent diagnosis of heart failure (HFrEF compared to HFpEF).

DETAILED DESCRIPTION:
The investigators will conduct a symptom assessment at study enrollment on cancer participants with a concurrent diagnosis of HF (HFrEF and HFpEF) using the MD Anderson Symptom Inventory- Heart Failure (MDASI-HF) and PROMIS Instruments (Fatigue, Dyspnea, and Sleep Disturbance).

The investigators will also describe and compare the health-related quality of life using the European Organization for Research and Training Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) and the measure of Quality of Life Short Form-12 (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Individuals with a concurrent solid tumor cancer diagnosis
* Not receiving active cancer treatment except for those on maintenance (i.e., Selective ER modulators (SERMs)[Tamoxifen], Aromatase inhibitors (Anastrozole, Letrozole, Exemestane), Ovarian suppression therapy (GnRH Agonists [Leuprolide], Androgen deprivation therapy for prostate cancer
* Completed cancer treatment at least 3 months and up to 3 years before study enrollment.

Therapy

* Able to read, speak and consent in English
* Ability to understand and the willingness to sign a written informed consent document
* Diagnosis of heart failure, confirmed by echocardiogram, MUGA, or cardiac catheterization
* Internet access via smart phone, tablet, a computer, or another device with the capacity to 1) download the Fitbit App and 2) complete electronic study assessments via REDCap.

Exclusion Criteria:

* Participants undergoing active cancer treatment.
* Inability to provide consent in the medical record, such as cognitively impaired individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will approach cancer participants with solid tumors and with a concurrent diagnosis of heart failure who are followed at MD Anderson for HF management. In fiscal year 2023, of the more than 20,000 hospital discharges, approximately 6% of those discharges have a concurrent diagnosis of heart failure. Investigators will enroll 100 participants who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Heart Failure | Through study completion, an average of 3 years
  The investigators will conduct a symptom assessment at study enrollment on cancer participants with a concurrent diagnosis of HF (HFrEF and HFpEF) using the MD Anderson Symptom Inventory- Heart Failure (MDASI-HF) and PROMIS Instruments (Fatigue, Dyspnea, and Sleep Disturbance).
Heart Failure | Through study completion, an average of 3 years
  The investigators will also describe and compare the health-related quality of life using the European Organization for Research and Training Quality- of-Life Questionnaire-Core 30 (EORTC QLQ-C30) and the Measure of Quality of Life Short Form-12 (SF-12).

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas of MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org